CLINICAL TRIAL: NCT02648555
Title: A Lifestyle Intervention to Improve in Vitro Fertilization Results
Acronym: W+D
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital dos Servidores do Estado do Rio de Janeiro (Other Government)
Collaborators: Gaffree & Guinle Universitary Hospital (Other)
Responsible Party: Principal Investigator, Silvia Hoirisch Clapauch, MD, PhD, Hospital dos Servidores do Estado do Rio de Janeiro
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Protocol W+D
Record Dates: First submitted 2016-01-04; First posted 2016-01-07 (Estimated); Last update posted 2016-01-07 (Estimated); Status verified 2016-01

CONDITIONS: Sterility; Placenta; Implantation; Risk Reduction Behavior; Lifestyle; Neonatal Hypoglycemia
MeSH Terms: conditions — Infertility; Risk Reduction Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard follow-up (controls) (No Intervention): Given that depressive disorders may increase the risk of spontaneous abortions, antidepressants will be not discontinued. However, expectant mothers on paroxetine or sertraline, which have been reported to increase the incidence of cardiac malformations, will be switched to fluoxetine.
- W+D protocol (lifestyle intervention) (Experimental): Daily walking and dietary recommendations. Expectant mothers on paroxetine or sertraline will be switched to fluoxetine
  Interventions: Behavioral: Daily walking; Behavioral: Dietary recommendations

INTERVENTIONS:
Behavioral: Daily walking — Participants will be instructed to walk briskly for >40 minutes, 7 days a week.
  Arms: W+D protocol (lifestyle intervention)
Behavioral: Dietary recommendations — Participants will be instructed to eat at least two daily servings of meat, poultry, fish (e.g. 2 g/kg) or other protein-rich food, starting at least one week before embryo transfer and continuing until delivery. They will be also recommended to avoid high-glycemic index meals (high-carbohydrate, low-fiber), such as snacks, candies, fiber-free juices, coconut water, and sugar-sweetened beverages, particularly carbonated soft drinks and sport drinks.
  Patients suffering from nausea usually do not tolerate solid food. As a result, fiber-free juices and sugar-sweetened beverages account of most of their caloric intake, which may cause non-adherence to the protocol. Women with nausea or vomiting will be treated with ondansetron.
  Arms: W+D protocol (lifestyle intervention)

SUMMARY:
Embryo adhesion and placentation depend on tissue plasminogen activator (tPA)-mediated activation of brain-derived neurotrophic factor, vascular endothelial growth factor and other growth factors, formation of hemidesmosomes, and degradation of extracellular matrix and basement membrane, either directly or by activating matrix metalloproteinases.

Since glucose and insulin stimulate release of a major tPA inhibitor by endothelial cells - plasminogen activator inhibitor (PAI)-1 - the investigators hypothesized that lifestyle interventions proven effective in maintaining glucose and insulin levels within the normal range would increase the take home baby rate in women undergoing assisted reproduction.

DETAILED DESCRIPTION:
Tissue plasminogen activator (tPA) has a well-known role in the coagulation pathway. tPA converts plasminogen to plasmin. Plasmin dissolves fibrin clots, thus limiting thrombus formation to the site of vascular injury.

In the extravascular compartment, tPA is a pivotal mediator of tissue formation and remodeling. Due to its proteolytic activity, tPA participates in processes as diverse as embryo adhesion, placental angiogenesis and vasculogenesis, and neuronal plasticity. Embryo adhesion and placentation, for example, depend on tPA-mediated activation of brain-derived neurotrophic factor, vascular endothelial growth factor and other growth factors, formation of hemidesmosomes, and degradation of extracellular matrix and basement membrane, either directly or by activating matrix metalloproteinases.

Assuming low tPA activity would impair both blood clot dissolution and placentation, the investigators postulated that patients with consecutive first-trimester abortions would have a high prevalence of severe dysmenorrhea, accompanied by the passage of large clots.

In 2011, the investigators assessed the prevalence of severe dysmenorrhea during early adolescence in two groups. The first one was made of women with ≥ 2 consecutive first-trimester abortions, and the other, of women with ≥ 2 living births, and no losses or preterm deliveries. Severe dysmenorrhea was defined as suprapubic menstrual cramp, intense enough to cause repeated absenteeism from school or fainting in the absence of analgesia. Early adolescents are unlikely to use contraceptives, or to have become pregnant, two situations that may reduce the pain. In this study, severe dysmenorrhea increased the chances of having consecutive first-trimester miscarriages by sevenfold (95% Confidence Interval: 3.4 to 14.1; p<0.001).

Since glucose and insulin stimulate release of a major tPA inhibitor by endothelial cells - plasminogen activator inhibitor (PAI)-1 - the investigators hypothesized that lifestyle interventions proven effective in maintaining glucose and insulin levels within the normal range would increase the take home baby rate in women undergoing assisted reproduction.

The protocol has already been tested at a Brazilian tertiary care center in women with unexplained consecutive first-trimester abortions, conceiving spontaneously. The objective of this study was to observe the impact of lifestyle interventions on the take home baby rate, and to observe if the intervention could reduce the prevalence of preeclampsia and neonatal hypoglycemia.

From 2011 to 2015, 480 patients aged 18 to 42 years with ≥ 2 consecutive first-trimester abortions documented by pathology or ultrasonography, were randomly assigned to protocol Walking and Diet (W+D) or to standard follow-up (controls). Women were enrolled independent of having had severe dysmenorrhea during adolescence. Patients assigned to protocol W+D were instructed to walk briskly for ≥ 40 minutes seven days a week. In addition, they were recommended to avoid high-carbohydrate meals such as snacks, candies, fiber-free juices, coconut water and sugar-sweetened beverages, and to eat two daily servings of meat, poultry, fish (e.g. 2 g/kg) or other protein-rich food, starting when they decided to get pregnant and continuing until delivery. Women with antiphospholipid antibodies, second- or third-trimester losses, multiple pregnancies, anatomical abnormalities that could increase the risk of first-trimester abortions, or any condition requiring a priori anticoagulation were excluded.

ELIGIBILITY:
Inclusion Criteria:

* women undergoing assisted reproduction

Exclusion Criteria:

1. liver failure, kidney failure or other conditions that prevent the patient from eating proteins.
2. multiple pregnancy.
3. paraplegia, hemiplegia, arthropathy and other conditions that prevent the participant from exercising.
4. participants lost to follow-up.
5. conditions that may strongly affect pregnancy results, such as a serious accident
6. participants assigned to non-intervention group following the recommendations given to intervention group.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 240 (Estimated)
Dates: Start 2016-05; Primary Completion 2018-05 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
The rate of viable pregnancies | two years

SECONDARY OUTCOMES:
The rate of fist trimester losses | four years
The rate of second and third trimester losses | four years
The rate of preeclampsia, eclampsia and HELLP syndrome | four years
Cramps or bleeding during the first trimester requiring progesterone | four years
The rate of prematurity | four years
The rate of intrauterine growth restriction | four years
Maternal weight gain | four years
The rate of gestational diabetes | four years
The rate of neonatal hypoglycemia | four years
The rate of neonatal hyperbilirubinemia requiring phototherapy | four years

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Hoirisch-Clapauch, MD, PhD, Principal Investigator — Hospital Federal dos Servidores do Estado, Ministry of Health
Locations (1):
- Hospital Federal dos Servidores do Estado, Ministry of Health, Rio de Janeiro, Rio de Janeiro, Brazil